CLINICAL TRIAL: NCT05819931
Title: Evaluation of the Effect of Respiratory Physiotherapy by Mechanical In-exsufflator on Respiratory Function in Patients with Amyotrophic Lateral Sclerosis: a Pilot Study
Brief Title: Breathing with Amyotrophic Lateral Sclerosis
Acronym: 2SLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC31/22/0411
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Mechanical In-Exsufflator; Physiotherapy; Cough; peak expiratory flow on cough
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Cough

STUDY DESIGN:
Intervention Model Description: before-after comparison of the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mechanical In-Exsufflator treatment (Experimental)
  Interventions: Device: Mechanical In-Exsufflator treatment

INTERVENTIONS:
Device: Mechanical In-Exsufflator treatment — The Mechanical In-Exsufflator (MIE) is a device that alternately inhales and exhales air and amplifies the respiratory cycles in flow and pressure. 15 breathing cycles (about 3 minutes) are recommended each day.
  Patients will practice the MIE daily independently and/or carried out by his physiotherapist (PT) during PT sessions.
  The MIE is prescribed by the neurologist or pulmonologist and is covered by social security in France. It is gifted by an external service provider.
  The Peak-Flow Cough is considered as the standardized score retaining the best of 3 consecutive measurements by Peak-Flow, a small portable device for personal use, which measures the maximum expiratory flow reached by the patient at the moment when the breath is most powerful.
  The patient is his own control. At baseline, the patient will be treated as usual. He will be asked to read the Peak-Flow Cough measures. The PT will also perform the Peak flow measurement at each patient visit.

SUMMARY:
The study aims to evaluate the effect of mechanical insufflator-exsufflator on the respiratory functions of Amyotrophic Lateral Sclerosis (ALS) patients evaluated via peak expiratory flow on cough (PEFC) measurements. The evolution of their PEFC is monitored to see if the curative management can have a positive impact on the latter.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a rare neurodegenerative pathology without curative treatment at present, the outcome is fatal after 3 to 5 years of evolution on average. The disease results in progressive paralysis of the muscles involved in voluntary motricity (progressive and intricate impairment of locomotor, phonation and swallowing capacities as well as ventilatory function). In France, the management of ALS is based on a diversified multidisciplinary follow-up (physiotherapy, speech therapy, occupational therapy, neuropsychology) in the ALS Reference Center in conjunction with the city care networks. It is centered on the evaluation, and the early compensation of the various symptoms, especially the respiratory problems.

Thus, this study aims to evaluate the effect of mechanical insufflator-exsufflator on the respiratory functions of these patients, evaluated via cough peak expiratory flow measurements (CPEF).

The study is conducted in collaboration with the physiotherapists of each patient enrolled, to evaluate the respiratory function by peak expiratory flow on cough (PEFC) after 4 weeks of treatment with Mechanical In-Exsufflator (MIE) (3 weekly sessions for two weeks, then one daily session for 2 weeks) in ALS patients presenting with a poorly effective cough (PEFC between 160 and 255 L/min) and having an indication of punctual MIE.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed ALS categorized as probable or certain according to the revised Awaji-Shima criteria [27].
* ALS of spinal, bulbar or respiratory forms
* Peak Flow measure between 160 and 255 L/min (recommendation of MIE in case of congestion, with the possibility of daily sessions)
* Patient who has not benefited from treatment by MIE in the past year (less than 10 sessions in total)
* Patient able to use the MIE and perform the collection, or having a caregiver able to help
* Patient receiving physiotherapist treatment greater than or equal to twice a week

Exclusion Criteria:

* Psychiatric (DSM-5) or cognitive disorders incompatible with participation in the study
* Contraindication to the use of an MIE (pneumothorax for example)
* Insufficient level in French for understanding the study and completing the questionnaires
* Current or past participation in another innovative research or care program relating to respiratory functions
* Emergency situation for which the MIE must be set up within less than a week

Exclusion during the study :

* Appearance of a serious contraindication to the practice of MIE during the study (for example rib fracture during a fall)
* Patient's physiotherapist refusing to do the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
cough peak expiratory flow evolution | 4 weeks post treatment initiation
  evolution of respiratory function by peak expiratory flow on cough (PEFC) after 4 weeks of treatment with Mechanical In-Exsufflator (3 weekly sessions for two weeks then one daily session for 2 weeks) in ALS patients presenting with a poorly effective cough (Cough Peak Expiratory Flow between 160 and 255) and having an indication of punctual MIE.
  Ratio between the PEFC 4 weeks post treatment initiation and PEFC at baseline can show decrease in respiratory function if <1 ; increase in respiratory functions if >1 and a conservation of respiratory function if = 1.
  A PEFC remaining within 10% of its initial value (rounded to the nearest ten) is considered unmodified

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lagarde, Principal Investigator — University Hospital, Toulouse
Locations (1):
- SLA Center - Purpan University Hospital Toulouse, FRANCE, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No